CLINICAL TRIAL: NCT03027635
Title: Tunnelated Peritoneal Catheter Versus Repeated Large Volume Paracentesis for Diuretic Resistant Ascites in Patients With Cirrhosis: An Investigator Initiated, Open, Parallel Arm Randomized Controlled Trial
Brief Title: PEriToneal Catheter Versus Repeated Paracentesis for Ascites in Cirrhosis
Acronym: PETRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and limited funding. The treatment intervention is instituted in clinical practice as and end-stage treatment option at hospitals in Denmark
Sponsor: Nina Kimer (Other)
Responsible Party: Sponsor-Investigator, Nina Kimer, MD, PhD, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PETRA21042016
Record Dates: First submitted 2016-12-13; First posted 2017-01-23 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Cirrhosis; Ascites Hepatic; Ascites (Non-Malignant)
Keywords: diuretic resistant ascites; Paracentesis; PleurX; Peritoneal tunnelated catheter
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Ciprofloxacin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PleurX (Experimental): The PleurX catheter is a tunnelated peritoneal catheter, designed for permanent placement in the peritoneal cavity. The catheter is placed by a physician under sterile conditions. Drainage of ascites is done using vacuum bottles connected to the catheter. This can be managed by a home nurse or the patient.
  Interventions: Device: PleurX, peritoneal tunnelated catheter; Drug: Ciprofloxacin 500Mg Tablet
- Large Volume Paracentesis (Active Comparator): Large volume paracentesis is performed in sterile technique, a small incision is made through the skin, and a catheter is inserted through muscle and peritoneum. After the procedure, the patient remains in hospital for observation until the fluid is drained.
  Interventions: Device: Large Volume Paracentesis; Drug: Ciprofloxacin 500Mg Tablet

INTERVENTIONS:
Device: PleurX, peritoneal tunnelated catheter — A permanent catheter
  Arms: PleurX
Device: Large Volume Paracentesis — Short time drainage
  Arms: Large Volume Paracentesis
Drug: Ciprofloxacin 500Mg Tablet — SBP prophylaxis

SUMMARY:
Insertion of a tunnelated peritoneal catheter (PleurX) allows repeated intermittent small volume fluid drainage at home. The treatment may improve the management of ascites and have a beneficial effect on the quality of life.

This study aims to evaluate the beneficial and harmful effects of the peritoneal catheter (PleurX) versus repeated large volume paracentesis for patients with cirrhosis and diuretic resistant ascites.

The trial is an investigator initiated, randomised, single blind, parallel arm, controlled trial.

Tunnelated peritoneal (PleurX) catheter versus large volume paracentesis. All patients will receive ciprofloxacin to prevent spontaneous bacterial peritonitis.

We will include 32 adult patients with cirrhosis Duration of trial 18 months. The total duration of follow up is six months. The primary outcome is paracentesis free survival.

DETAILED DESCRIPTION:
Ten percent of patients with cirrhosis develop ascites. In 90% of patients, ascites can be treated with diuretics. The management of the remaining 10% with diuretic resistant ascites is challenging. Symptoms including abdominal pain, dyspnoea, nausea, vomiting, and anorexia have a detrimental impact on the quality of life. Repeated large volume paracentesis provides only temporary improvement of symptoms.

Insertion of a tunnelated peritoneal catheter (PleurX) allows repeated intermittent small volume fluid drainage at home. The treatment may improve the management of ascites and have a beneficial effect on the quality of life.

To evaluate the beneficial and harmful effects of the peritoneal catheter (PleurX) versus repeated large volume paracentesis for patients with cirrhosis and diuretic resistant ascites.

Investigator initiated, randomised, single blind, parallel arm, controlled trial.

Due to the nature of the intervention and the primary outcome measure, Investigators are unable to conduct the trial with blinding of the patients, the investigators or use blinded outcome assessment.

Tunnelated peritoneal (PleurX) catheter versus large volume paracentesis. All patients will receive ciprofloxacin to prevent spontaneous bacterial peritonitis.

The study investigators will include 32 adult patients with cirrhosis of any aetiology and diuretic resistant ascites.

Gastrounit, Hvidovre University Hospital, Department of Gastroenterology and Hepatology, Odense University Hospital, Department of Gastroenterology and Hepatology, Aarhus University Hospital, and Centre for Hepatology, UCL Institute for Liver and Digestive Health, Royal Free Campus, University College London, UK 18 months. The total duration of follow up is six months. The primary outcome is paracentesis free survival. Secondary outcomes include cumulative number of paracentesis, cirrhosis-related complications, safety, quality of life, changes in metabolic and nutritional parameters, circulatory dysfunction, renal function, cardiac output, neuro-humoral changes.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any aetiology
* Diuretic resistant ascites defined as i) an inability to mobilise ascites (minimal or no weight loss) despite administration with the maximum tolerable doses of oral diuretics or a daily dose of spironolactone 400 mg and re-accumulation of fluid after therapeutic paracentesis within two weeks or ii) diuretic-related complications including (but not limited to) azotemia, hepatic encephalopathy, or progressive electrolyte imbalances
* Able to read and understand Danish
* Signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female of any age
* Age at least 18 years
* Expected survival at least three months.

Exclusion Criteria:

* Participants eligible and listed for TIPS
* Serum creatinine levels above 135 umol/L
* Overt hepatic encephalopathy in the two weeks before randomization
* Ascites due to other causes than cirrhosis such as: malignant disease, congestive heart failure, end-stage renal disease, pancreatitis, or Budd-Chiari (hepatic vein thrombosis), or chylous ascites
* Ongoing intra-abdominal infection (peritonitis) or active systemic or local infections, such as urinary tract infection or pneumonia
* Participation in a clinical study that may interfere with participation in this study;
* Evidence of extensive ascites loculation
* Coagulopathy
* Variceal bleeding within two weeks before randomisation
* Intraabdominal surgery within four months before randomisation
* Spontaneous bacterial peritonitis (neutrophil count>250/µl within 24 hours of randomization)
* Patients with an increased risk of procedure related complications as judged by the primary healthcare provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Time to first paracentesis | 18 months

SECONDARY OUTCOMES:
Adverse events | 18 months
  Number of AEs in groups
Nutritional Status | 18 months
  Indirect calorimetry
Renal function | 18 months
  glomerular filtration rate
Cardiac Output | 18 months
  cardiac output

CONTACTS AND LOCATIONS:
Locations (1):
- Gastro Unit, medical Division, University Hospital Hvidovre, Hvidovre, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Due to Danish Legislation only anonymized data may be available upon request